CLINICAL TRIAL: NCT06614595
Title: Transfusion in Lower Risk MDS Patients: Predictors of Adequacy of Transfusion and Quality of Life Changes
Brief Title: Transfusion in Lower Risk MDS Patients: Predictors of Adequacy of Transfusion and Quality of Life in Lower Risk MDS
Acronym: MDS-QUAL
Status: Recruiting | Type: Observational
Sponsor: Fundación para la Investigación Biosanitaria del Principado de Asturias (Other)
Collaborators: Hospital Universitario Central de Asturias (Other)
Responsible Party: Principal Investigator, Teresa Bernal del Castillo, Principal Investigator, MD, PHD, Fundación para la Investigación Biosanitaria del Principado de Asturias
Other Study IDs: 2024.244
Record Dates: First submitted 2024-09-24; First posted 2024-09-26 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Low Risk Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndromes; Red blood cell transfusion; Quality of life
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and plasma for cytokine analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study to evaluate changes in quality of life (QoL) in patients diagnosed with low risk MDS who are red blood cell (abc) transfusion dependent.

Changes in QoL will be correlated with patient cardiorespiratory function. Cardiac biomarkers and plasma cytokines will also be evaluated.

DETAILED DESCRIPTION:
At inclusion and before red blood cell (rbc) transfusion, patients cardiorespiratory function will be evaluated with an ergospirometer

Likewise, before and after rbc transfusion, patients will be asked to complete the QUALMS, a QoL instrument which will be supplied by Dr. Gregory Abel at Dana-Farber in the U.S., who led its development team.

Before and after rbc transfusion, hemoglobin, pretrasfusional hemoglobin, pre and post cardiac biomarkers troponin and NTproBNP will be collect.Pre and post serum and plasma will also be collected for cytokine analysis.

ELIGIBILITY:
Subjects must meet all of the following inclusion criteria:

1. They must be able to understand the study procedures, comply with them, and consent in writing prior to any specific study procedure.
2. Must be able to understand the study procedures, comply with them, and give written informed consent prior to any study-specific procedure.
3. Adult subjects ≥ 18 years of age with a diagnosis of myelodysplastic syndrome.
4. Very low, low or intermediate IPSS-R risk category.
5. Subject requires are red blood cell transfusion dependent with the following criteria: requires an average of 2 to 6 units of CH on average over an 8-week period.
6. ECOG 0-3.

Exclusion criteria

1. Subject undergoing any of the following treatments: azacitidine, decitabine, venetoclax, cytotoxic chemotherapy, radiotherapy, arsenic trioxide, interferon or interleukin.
2. High or very high IPSS-R risk category.
3. Subject diagnosed with any active neoplasm except:

   * epidermoid or basal cell carcinoma,
   * carcinoma in situ of the uterine cervix
   * Carcinoma in situ of the breast
4. Subjects with a score on the New York Heart Association Scale IV.
5. Subjects with major surgery within 8 weeks prior to study inclusion. Subjects must have fully recovered from any previous surgery prior to inclusion in the study.
6. Subject with known clinically significant anaemia due to iron, vitamin B12 or folate deficiencies or autoimmune or hereditary haemolytic anaemia or uncontrolled hypothyroidism or known clinically significant haemorrhage or sequestration or subject with drug induced anaemia.
7. New onset or uncontrolled seizures.
8. Subjects with uncontrolled systemic fungal, bacterial or viral infections (defined as ongoing signs or symptoms related to the infection without improvement despite appropriate antibiotics or antimicrobial therapy).
9. Pregnant or breastfeeding women.
10. The subject has any condition, including the presence of laboratory abnormalities that would place the subject at unacceptable risk if he/she were to participate in the study.
11. The subject has any condition or receives concomitant medication that confounds the ability to interpret the study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lower-risk Myelodysplastic syndrome patients, red blood cell transfusion dependent
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Prediction of Quality of Life (QoL) improvement, assessed by an increase in 5 points or more in the QUALMs scale | We expect to obtain results in one year from the beginning of the study
  To design a score that help to identify which patients benefit from red blood cell Transfusion in terms of QoL improvement

SECONDARY OUTCOMES:
Changes in QoL before and after transfusion | QoL will be asses the day of transfusion and seven days after
  QoL will be assessed with QUALMS instrument, The QUALMS is being supplied by Dr. Gregory Abel at Dana-Farber in the U.S., who led its development team. He will collaborate and assist in the interpretation of the HRQoL results.

OTHER OUTCOMES:
Troponin and NTproBNP as predictors for QoL improvement | Troponin and NTproBNP will be analyzed the day of transfusion and seven days after
  To evaluate the utility of serum pretransfusional troponine and NTPROBNP as cardiac biomarkers to identify those patients whose QoL improves after the rbc transfusion
Cardiorespiratory function | Ergospirometry will be performed at the inclusion in the study
  To evaluate the utility of oxygen consumption measured by ergospirometry to evalaute cardiorespiratory function and as a predictor of QoL improvement after rbc transfusion
Cytokines | Cytokines will be analyzed before abc transfusion and seven days after it
  To analyze changes in pro and anti-inflammatory cytokines before and after rbc transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abel GA, Efficace F, Buckstein RJ, Tinsley S, Jurcic JG, Martins Y, Steensma DP, Watts CD, Raza A, Lee SJ, List AF, Klaassen RJ. Prospective international validation of the Quality of Life in Myelodysplasia Scale (QUALMS). Haematologica. 2016 Jun;101(6):781-8. doi: 10.3324/haematol.2015.140335. Epub 2016 Mar 4. PMID 26944474
- [Background] Abel GA, Klepin HD, Magnavita ES, Jaung T, Lu W, Shallis RM, Hantel A, Bahl NE, Dellinger-Johnson R, Winer ES, Zeidan AM. Peri-transfusion quality-of-life assessment for patients with myelodysplastic syndromes. Transfusion. 2021 Oct;61(10):2830-2836. doi: 10.1111/trf.16584. Epub 2021 Jul 12. PMID 34251040